CLINICAL TRIAL: NCT00464113
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL228 Administered Intravenously to Subjects With Chronic Myeloid Leukemia (CML) or Philadelphia-Chromosome-Positive Acute Lymphocytic Leukemia (Ph+ ALL)
Brief Title: Study of XL228 in Subjects With Chronic Myeloid Leukemia or Philadelphia-Chromosome-Positive Acute Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL228-001
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Myeloid Leukemia; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive
Keywords: Myeloid Leukemia; Lymphocytic Leukemia; Ph+ ALL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid; Leukemia, Lymphoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): once-weekly dosing
  Interventions: Drug: XL228
- 2 (Experimental): twice-weekly dosing
  Interventions: Drug: XL228

INTERVENTIONS:
Drug: XL228 — 1-hour IV infusion

SUMMARY:
The purpose of this study is to determine the safest dose of the BCR-ABL inhibitor XL228, how often it should be taken, and how well people with leukemia tolerate XL228.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a confirmed pathologic diagnosis as evidenced by the presence of the BCR-Abl translocation [t(9;22)] by fluorescence in situ hybridization (FISH), cytogenetics, or quantitative polymerase chain reaction (QPCR) of one of the following:

   1. CML

      * Chronic phase (CP)
      * Accelerated phase (AP)
      * Blast phase (BP) OR
   2. Ph+ ALL
2. The subject has one of the following:

   * Known T315I Abl mutation
   * Known resistance to or intolerance of imatinib and dasatinib
   * At least one prior anti-leukemia therapy, including, but not limited to, interferon, imatinib, or dasatinib
3. The subject is at least 18 years old.
4. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
5. The subject has adequate organ function.
6. The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
7. Sexually active subjects must use an accepted method of contraception during the course of the study.
8. Female subjects of childbearing potential must have a negative pregnancy test at enrollment.

Exclusion Criteria:

1. The subject has received interferon, imatinib, or dasatinib within 7 days of the first dose of XL228.
2. The subject has received an investigational agent or radiotherapy within 28 days of the first dose of XL228.
3. The subject has received immunosuppressive therapy (eg, cyclosporine, steroids, tacrolimus for graft-versus-host disease [GVHD]) within 28 days prior to the first dose of XL228.
4. The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤1 from toxicities related to peripheral stem cell or bone marrow transplant.
5. The subject has not recovered to CTCAE v3.0 Grade ≤1 from adverse events (AEs) due to investigational drugs or other medications.
6. The subject has known allergy or hypersensitivity to any component of the investigational drug product.
7. The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. The subject is pregnant or breastfeeding.
9. The subject is known to be positive for the human immunodeficiency virus (HIV).
10. The subject has an inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of once-weekly and/or twice-weekly 1-hour intravenous (IV) infusion of XL228 | Assessed at periodic visits

SECONDARY OUTCOMES:
Evaluate plasma pharmacokinetics and estimate renal elimination of once-weekly and twice-weekly 1-hour IV infusion of XL228 | Assessed at periodic visits
Exploratory Outcomes: Evaluate hematologic and cytogenetic response and pharmacodynamic correlates of XL228 activity | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA School of Medicine, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Georgetown University Medical Center, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Michigan Health System, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas